CLINICAL TRIAL: NCT06319729
Title: The Efficacy and Safety of a Chinese Herbal Medicine for the Constipation-predominant Irritable Bowel Syndrome (IBS-C): a Double-blinded, Placebo-controlled, Randomized Pilot Clinical Trial
Brief Title: A Chinese Herbal Medicine for IBS-C
Acronym: CDD2105RCT1
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, ZhaoXiang Bian, Prof., Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REC/22-23/0659
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Constipation-predominant Irritable Bowel Syndrome
Keywords: Chinese Herbal Medicine; IBS-C

STUDY DESIGN:
Intervention Model Description: A double-blind, placebo-controlled randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All the study drugs and placebo should be in the same package with the same drug appearance and blinded according to the randomized numbers of the subgroups. The specific blinding method is set as follows: the study drugs and placebo are uniformly packaged and numbered according to the corresponding randomized group results. One copy of the blinding letter in duplicate is sent with the test drug to the project leader of the test center for storage, and the other copy is kept by the pharmacy until the end of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): During the 4-week intervention, participants are required to consume 4.7g of CDD-2105 granule (a Chinese herbal medicine formula containing four granular herbs) twice per day.
  Interventions: Drug: CDD-2105
- Placebo group (Placebo Comparator): During the 4-week intervention, participants are required to consume 4.7g of placebo twice per day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CDD-2105 — A Chinese herbal medicine formula containing four granular herbs.
  Arms: Treatment group
Drug: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
This double-blind, placebo-controlled randomized pilot clinical trial will test the hypothesis that granules of CDD-2105, a Chinese herbal medicine formula, will have efficacy in alleviating constipation and abdominal pain in individuals with IBS-C. Participants (n=78) will be randomly assigned to the treatment or placebo group in a 1:1 ratio, followed by 4 weeks of intervention and 4 weeks of follow-up.

DETAILED DESCRIPTION:
This double-blind, placebo-controlled randomized pilot clinical trial will test the hypothesis that granules of CDD-2105, a Chinese herbal medicine formula, will have efficacy in alleviating constipation and abdominal pain in individuals with IBS-C. Participants (n=78) will be randomly assigned to the treatment or placebo group in a 1:1 ratio, followed by 4 weeks of intervention and 4 weeks of follow-up.Primary Objective: To determine the efficacy and safety of CDD-2105 granules for treating IBS-C.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years adults
* Fulfill the clinically diagnosed with IBS-C based on the ROME IV criteria
* Abdominal pain intensity: weekly average of the worst daily (in the past 24 hours) abdominal pain score of ≥3.0 on a 0 to 10 point scale (based on the 2-week E-diary in screening)
* CSBM ≤ 2 times/week (based on the 2-week E-diary in screening)
* Understand and be able to follow written and oral instructions in Chinese
* Provide informed consent
* Able to use and complete 2-week E-diary for screening

Exclusion Criteria:

* Drug-induced or secondary causes of constipation
* Use of medications and/or supplements that may confound the study outcomes (including but not limited to antibiotics, steroid, analgesic drug, neuromodulator, prebiotics, symbiotics, or probiotics)
* Clinically significant colonoscopy or sigmoidoscopy examination findings after the onset of symptoms for patients who (1) is ≥50 years old; and/or (2) has family risk of colon-rectal cancer or familial polyposis syndromes; and/or (3) has alarm symptoms within 6 months before screening (unintentional weight loss: >10% in 3 months, blood in the stools not caused by hemorrhoids or anal fissures, fever of unknown origin, anemia)
* Clinically significant laboratory or imaging findings within 6 months before screening
* Recent history of mushy or watery stools within one month
* Allergic to Chinese herbal medicine or G6PD
* Abdominal surgeries within the past year (except laparoscopic appendectomy)
* Pregnancy, breastfeeding or plan to become pregnant with the study timeframe
* Any disease(s), condition(s) or habit(s) deemed by the investigators that would compromise the individual's ability to complete the study, e.g. serious psychiatric conditions, at the discretion of the investigators
* Any disease(s), condition(s) or habit(s) deemed by the investigators that would prevent participation in the study, e.g. participation in past or active clinical research, at the discretion of the investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-03-25 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Abdominal Pain Responder Rate | from baseline to Week 4
  An abdominal pain responder is a patient who meets the abdominal pain weekly responder criterion (i.e., an improvement of ≥30% from the baseline weekly average of the worst abdominal pain in the past 24 hours score to the weekly average during the intervention, in at least 2 out of 4 weeks). Abdominal pain at its worst (in the last 24 hours) is assessed daily by participants on an 11-point numerical rating scale where 0 represents no abdominal pain and 10 represents very severe abdominal pain. Baseline of weekly abdominal pain will be the average between Week -2 and Week 0.
Complete Spontaneous Bowel Movement (CSBM) Responder Rate | from baseline to Week 4
  A CSBM responder is defined as a patient who meets the CSBM responder criterion (i.e., a mean increase of CSBM≥1/week compared with CSBM at baseline, in at least 2 out of 4 weeks). A spontaneous bowel movement (SBM) is defined as a bowel movement without laxative use in the preceding 24 hours. A CSBM is defined as a SBM that is associated with a sense of complete evacuation. Baseline of weekly CSBM will be the average between Week -2 and Week 0.

SECONDARY OUTCOMES:
Change in the weekly average self-assessed daily maximum abdominal pain scores (0-10) | from baseline to Week 4
  weekly average self-assessed daily maximum abdominal pain scores (0-10)
Change in the number of days of abdominal pain per week | from baseline to Week 4
  weekly number of days of abdominal pain
Change in the average weekly Complete Spontaneous Bowel Movement (CSBM) frequency | from baseline to Week 4
  weekly Complete Spontaneous Bowel Movement (CSBM) frequency
Change in the average weekly Spontaneous Bowel Movement (SBM) frequency | from baseline to Week 4
  weekly Spontaneous Bowel Movement (SBM)
Change in the score of Irritable Bowel Syndrome-Severity of Symptoms (IBS-SSS) questionnaire | from baseline to Week 4
  Irritable Bowel Syndrome-Severity of Symptoms (IBS-SSS), 0-500, Mild, moderate and severe cases are indicated by a score of 75 to 175, 175 to 300 and greater than 300, respectively.
Change in the score of Patient Assessment of Constipation-Symptoms (PAC-SYM) | from baseline to Week 4
  Patient Assessment of Constipation-Symptoms (PAC-SYM), It is five - grade (0-4)likert scale. The high scores indicate worsening severity of symptoms.
Change in the score of Patient Assessment of Constipation Quality of Life (PAC-QoL) questionnaire | from baseline to Week 4
  Patient Assessment of Constipation Quality of Life (PAC-QoL). The PAC-QOL questionnaire is subcategorized to 4 items on physical discomfort, 8 items on psychosocial discomfort, 5 items on treatment satisfaction, and finally 11 items on worries and discomfort. Response choice is a Likert scale from 0 to 4. Higher scores mean higher negative effects on quality of life.
Safety: number of adverse events | from baseline to Week 4
  Assessed by number of adverse events or side effects
Safety: the level of liver function (ALT, AST, AKP, GGT, TBIL, DBIL) and renal function (blood urea nitrogen, creatinine) | from baseline to Week 4
  Assessed by liver and renal related index in blood samples

IPD SHARING:
Plan to Share IPD: Yes
The protocol, SAP, and de-identified data will be shared upon the researchers' request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months
Access Criteria: researchers' request